CLINICAL TRIAL: NCT06462235
Title: A PHASE 2A, 2-PART, OPEN-LABEL, NON-RANDOMIZED, MULTICENTER, SINGLE AND MULTIPLE DOSE TRIAL TO EVALUATE PHARMACOKINETICS, SAFETY AND TOLERABILITY OF AZTREONAM AND AVIBACTAM ± METRONIDAZOLE IN NEONATES AND INFANTS FROM BIRTH TO LESS THAN 9 MONTHS OF AGE WITH SUSPECTED OR CONFIRMED INFECTIONS DUE TO GRAM-NEGATIVE PATHOGENS REQUIRING INTRAVENOUS ANTIBIOTIC TREATMENT
Brief Title: A Study to Learn About the Study Medicine Aztreonam-Avibactam (ATM-AVI) in Infants and Newborns Admitted in Hospitals With Bacterial Infection (CHERISH)
Acronym: CHERISH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C3601010; 2023-507757-15-00 (Registry Identifier: CTIS (EU)); CHERISH (Other: Alias Study Number)
Record Dates: First submitted 2024-05-28; First posted 2024-06-17 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Gram-negative Bacterial Infection
Keywords: gram-negative; aztreonam-avibactam; neonate; infant
MeSH Terms: conditions — Gram-Negative Bacterial Infections

STUDY DESIGN:
Intervention Model Description: Non-randomized, 2-part with four age cohorts in each part
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A, Cohorts 1-4 (Experimental): Single dose pharmacokinetics.
  Interventions: Drug: Part A: ATM-AVI Single Dose, Cohorts 1-4
- Part B, Cohorts 1-4 (Experimental): Multi-dose pharmacokinetics and treatment
  Interventions: Drug: Part B: Multiple-dose ATM-AVI, Cohorts 1-4

INTERVENTIONS:
Drug: Part A: ATM-AVI Single Dose, Cohorts 1-4 — Single intravenous infusion of aztreonam-avibactam over 3 hours to assess pharmacokinetics, safety, and toleration.
  Arms: Part A, Cohorts 1-4
Drug: Part B: Multiple-dose ATM-AVI, Cohorts 1-4 — Multiple intravenous infusions of aztreonam-avibactam over 3 hours, repeated every 6-8 hours up to 14 days to assess pharmacokinetics, safety, toleration, and efficacy.
  Arms: Part B, Cohorts 1-4

SUMMARY:
The purpose of this study is to learn about the safety and effects of ATM-AVI for the possible treatment of infections caused by a type of bacteria called gram-negative bacteria.

The study medicine is a combination of an antibiotic, aztreonam (ATM), and another medicine, avibactam (AVI), which is used to help stop bacteria from being resistant to antibiotics. Antibiotics are medicines that fights bacteria and infections.

The study will include newborns and infants up to 9 months of age who are admitted in the hospital.

The study is conducted in 2 parts: Part A and Part B.

In Part A, all participants will receive a single intravenous (injected directly into a vein) infusion of ATM-AVI. This is to study the safety and effects of a single amount.

In Part B, all participants will receive multiple intravenous infusions of ATM-AVI as treatment for a possible or confirmed infection with gram-negative bacteria.

DETAILED DESCRIPTION:
This is a 2-part Phase 2a, non-randomized, multicenter, open-label, single and multi-dose study to assess pharmacokinetics (PK), safety, and tolerability of ATM-AVI in hospitalized neonates and infants aged birth, including preterm birth, to <9 months. A total of 48 participants will be enrolled in 4 age cohorts of 12 each, 6 Part A and 6 Part B. Part A will begin enrolling before Part B and no infant may participate in both parts. Cohort 1 will include full term infants age ≥13 weeks to <39 weeks and preterm infants postmenstrual age ≥50 weeks to <75 weeks. Cohort 2 will include full term infants age ≥28 weeks to <13 weeks and preterm infants postmenstrual age ≥40 weeks to <50 weeks and ≥28 days of age. Cohort 3 will include full term infants age birth to <28 days. Cohort 4 will include preterm infants age birth to <28 days or postmenstrual age <40 weeks.

Participants in Part A must be hospitalized and receiving intravenous antibiotic treatment for a suspected or confirmed bacterial infection. Participants will receive a single 3 hour intravenous infusion of ATM-AVI and have 3 ATM-AVI blood level assessments during and up to 5 hour after the infusion. Participants will be observed for 48 hours following the infusion to assess safety and toleration and will have a final follow-up safety assessment which may be conducted by telephone 4-5 weeks following the infusion. The single infusion of ATM-AVI is administered to assess the safety, tolerability, and pharmacokinetics of a single dose of ATM-AVI and is not intended as treatment for the bacterial infection. The total duration of study participation in Part A is expected to be 5 weeks through the end of the final safety follow-up.

Participants in Part B must be hospitalized with suspected or confirmed aerobic gram-negative bacterial infection requiring intravenous antibacterial therapy. Part B participants will receive multiple 3 hour intravenous infusions of ATM-AVI every 6 hour (8 hours for preterm infants) for 3-14 days as treatment for their bacterial infection and to assess ATM-AVI pharmacokinetics, safety, tolerability, and efficacy. Participants with complicated intra-abdominal infection (cIAI) will also receive intravenous metronidazole and all participants will have the option to receive other intravenous antibiotic treatment for gram-positive bacteria, as appropriate. Participants who have a good clinical response after 72 hours of intravenous ATM-AVI treatment may be switched to a different orally administered antibiotic, if clinically appropriate. Part B participants will have a total of 5 ATM-AVI blood level assessments over the first 2 or more days following the start of ATM-AVI infusions and will have their clinical response assessed at the End of Treatment (intravenous and oral, if applicable), and at a Test-of-Cure (TOC) evaluation 7 to 14 days after the last antibiotic treatment (intravenous or oral). A final safety assessment which may be conducted by telephone will occur 4-5 weeks after the last dose of ATM-AVI. The total duration of study participation in Part B is expected to be up to 7 weeks through the end of the final safety follow-up.

Additional safety monitoring will be provided by an independent external Data Monitoring Committee (DMC). Enrollment for the study will begin with Part A, single dose, cohorts 1-3. Part A Cohort 4 (preterm neonates) will commence enrollment after sponsor and DMC review of plasma drug levels and safety for a least 2 participants in Part A Cohort 3 and review of ATM-AVI safety and tolerability for all participants enrolled at that time. Enrollment in the multidose Part B cohorts will be delayed until preliminary information is obtained regarding ATM-AVI multidose safety, tolerability, and drug levels for the participants 9 months to 2 years of age in the separate ongoing ATM-AVI pediatric study C3601008 [NCT05639647].

ELIGIBILITY:
Inclusion Criteria

Participants must meet the following key inclusion criteria to be eligible for enrollment into the study:

1. Hospitalized with age from birth <9 months, including preterm birth
2. Part A: Receiving IV antibiotics for treatment of suspected or confirmed bacterial infection, including but not limited to cIAI, cUTI, HAP/VAP, BSI, or sepsis.
3. Part B: Suspected or confirmed gram-negative bacterial infection requiring IV antibiotics, including but not limited to cIAI, cUTI, HAP/VAP, BSI, or sepsis.

Participants with any of the following characteristics/conditions will be excluded:

1. Received any other investigational medicinal product within the longer of 30 days or 5 half-lives before enrollment.
2. Any medical or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
3. Severe renal impairment or known significant renal disease, as evidenced by elevated serum creatinine at screening, or urinary output <0.5 mL/kg/h for 6 consecutive hours or requirement for dialysis.
4. Part B Only: Received >24 hours of systemic antibiotic treatment for gram-negative organisms at time of enrollment, unless documented treatment failure or lack of improvement in at least one objective sign or symptom of infection after ≥48 hours of antibiotics.

Max Age: 39 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2027-12-02 (Estimated); Study Completion 2027-12-02 (Estimated)

PRIMARY OUTCOMES:
Maximum Predicted Plasma Concentration (Cmax) of ATM and AVI | Up to Day 15
  Cmax is the maximum plasma concentration of ATM and AVI as population pharmacokinetic (popPK) analysis predicts.
Area under the Concentration-Time Curve (AUC) of ATM-AVI | Up to Day 15
  AUC is a measure of the plasma concentration of ATM and AVI overtime as popPK analysis predicts.
Plasma Elimination Half-Life (t1/2) | Up to Day 15
  Half-life is the time measured for the plasma concentration of ATM and AVI to decrease by one half as popPK analysis predicts.
Apparent Clearance (CL) | Up to Day 15
  ATM and AVI clearance is a quantitative measure of the rate at which ATM and AVI are removed from the blood (rate at which ATM and AVI are metabolized or eliminated by normal biological processes). Clearance obtained after intravenous infusion dose (apparent clearance) is influenced by the fraction of the dose absorbed.
Plasma concentrations of ATM and AVI by nominal sampling time | Up to Day 15
  Plasma concentrations of ATM and AVI on Day 1 and at steady state (Day 2 or later) will be summarized by the nominal sampling time using descriptive statistics (eg number, mean, standard deviation).
Proportion of Participants reporting Adverse Events (AE) | Baseline up to Day 50
  Proportion of participant AE reports of vital signs, physical examinations, and clinical laboratory tests overall and by age cohort. For each AE the last assessment made prior to the first dose of study drug will be defined as the baseline.
Proportion of Participants reporting Serious Adverse Events (SAE) | Baseline up to Day 50
  Proportion of participant SAE reports of vital signs, physical examinations, and clinical laboratory tests overall and by age cohort. For each SAE the last assessment made prior to the first dose of study drug will be defined as the baseline.
Proportion of Participants reporting AEs leading to discontinuation of study drug | Baseline up to Day 50
  Proportion of Participants reporting AEs leading to discontinuation of study drug from baseline. For each discontinuation the last assessment made prior to the first dose of study drug will be defined as the baseline.
Proportion of Participants reporting AEs resulting in death | Baseline up to Day 50
  Proportion of Participants reporting AE resulting in death from baseline. For each death the last assessment made prior to the first dose of study drug will be defined as the baseline.
Proportion of Participants reporting liver injury and acute kidney injury | Baseline up to Day 50
  Proportion of Participants reporting liver injury and acute kidney injury from baseline. For each report of liver and acute kidney injury the last assessment made prior to the first dose of study drug will be defined as the baseline.

SECONDARY OUTCOMES:
Part B: Proportion of participants with each clinical outcome and with a favorable clinical outcome at end of IV study treatment (EOIV) | Up to 15 days after start of IV study treatment
  Clinical Cure is defined baseline signs and symptoms improved such that no further antimicrobial treatment is required for an aerobic gram-negative baseline infection. Participants who receive treatment for gram-positive organisms or adjunctive therapy for Pseudomonas aeruginosa, as allowed per protocol, can still have a response of cure. Clinical improvement is defined as baseline signs and symptoms sufficiently improved to allow switching to an oral antibiotic treatment. A favorable outcome is clinical cure or clinical improvement. Failure is defined as a requirement for further antibiotic treatment, including following premature discontinuation due to an adverse event, or death after receiving at least 48 hours of treatment. Indeterminant is defined as data not available for evaluation of efficacy for any reason.
Part B: Proportion of participants with each clinical outcome and with a favorable clinical outcome at end of treatment (EOT) | Within 48 hours after last dose of oral switch treatment
  EOT is only applicable for participants switched to an oral antibiotic treatment. Possible outcomes are cure, failure, or indeterminant.
Part B: Proportion of participants with each clinical outcome and with a favorable clinical outcome at test of cure (TOC) | 7-14 days after the last study treatment
  Possible outcomes are cure, failure, or indeterminant.
Part B: Proportion of participants with a favorable microbiological response at TOC | 7-14 days after the last study treatment
  A favorable response is eradication or presumed eradication. Eradication is absence of the causative pathogen from an appropriately obtained specimen at the site of infection. Presumed eradication is when a repeat culture was not performed and the clinical response is cure.
Part B: Counts and proportions of pathogens with each per-pathogen microbiological response at EOIV/EOT | Up to 15 days after start of IV study treatment
  Possible outcomes are eradication, presumed eradication, persistence, presumed persistence or indeterminate. Presumed eradication/persistence based on repeat culture not performed and clinical outcome of cure/failure. Persistence is the causative pathogen is still present from an appropriately obtained specimen at the site of the infection. Indeterminant includes participant lost to follow-up or death after receiving less than 48 hours of study treatment.
Part B: Counts and proportions of pathogens with each per-pathogen microbiological response at TOC | 7-14 days after the last study treatment
  Possible outcomes are eradication, presumed eradication, persistence, presumed persistence or indeterminate.
Part B: Counts and proportions of participants with emergent infections (new infections or superinfections) during the study | Through study completion, up to Day 50
  Superinfection is defined as emergence of a new pathogen associated with worsening signs and symptoms of infection and a requirement for additional antibiotics during the period up to and including EOIV/EOT. New infection is defined as emergence of a new pathogen associated with worsening signs and symptoms of infection and a requirement for additional antibiotics during the period after EOIV/EOT.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (28):
- United States (13):
  - Children's Hospital of Orange County Southwest Tower, Orange, California
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Norton Children's Hospital, Louisville, Kentucky
  - Novak Center for Children's Health, Louisville, Kentucky
  - University of Louisville, Norton Children's Research Institute, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Bristol Myers Squibb Children's Hospital at Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers University, New Brunswick, New Jersey
  - Duke University - Main Hospital and Clinics, Durham, North Carolina
  - Memorial Hermann Hospital - Texas Medical Center, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
- Argentina (4):
  - Sanatorio Sagrado Corazón, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Clinica Del Niño Y La Madre, Mar del Plata, Buenos Aires
  - Clinica Privada del Sol S.A, Córdoba, Córdoba Province
  - Hospital del Niño Jesús, San Miguel de Tucumán, Tucumán Province
- India (4):
  - Nirmal Hospital Pvt Ltd., Surat, Gujarat
  - RajaRajeswari Medical College and Hospital, Bengaluru, Karnataka
  - Medanta Hospital Lucknow, Lucknow, Uttar Pradesh
  - Institute of Child Health, Kolkata, West Bengal
- Israel (2):
  - Schneider Children's Medical Center, Petah Tikva, Central District
  - Rambam Health Care Campus, Haifa, Northern District
- Taiwan (5):
  - Hsinchu Municipal Mackay Children's Hospital, Hsinchu, Hsinchu
  - Hualien Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Hualien City, Hualien
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3601010